CLINICAL TRIAL: NCT05224583
Title: Prevalence of BK Viremia in Simultaneous Liver-Kidney Transplant Recipients: A Retrospective Single-Center Review
Brief Title: Prevalence of BK Viremia in Simultaneous Liver-Kidney Transplant
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 052.MTP.2021.D
Record Dates: First submitted 2022-02-03; First posted 2022-02-04 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Polyomavirus Infections; BK Viremia; Liver Transplant Infection; Kidney Transplant Infection
MeSH Terms: conditions — Polyomavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Simultaneous Liver-Kidney Transplant patients population at MDMC: Consecutive SLK transplant recipients who were transplanted at MDMC over a 6-year period (2015 to 2020).
  Interventions: Procedure: Simultaneous Liver-Kidney Transplant

INTERVENTIONS:
Procedure: Simultaneous Liver-Kidney Transplant — Simultaneous Liver-Kidney Transplant

SUMMARY:
The human BK polyomavirus is a significant risk factor for renal transplant dysfunction and allograft loss. The prevalence of BK viremia (BKV) following kidney transplantation is estimated to be 10-20%.

DETAILED DESCRIPTION:
The human BK polyomavirus is a significant risk factor for renal transplant dysfunction and allograft loss. The prevalence of BK viremia (BKV) following kidney transplantation is estimated to be 10-20%. Immunosuppression reduction is the management cornerstone for BKV and has been shown to be effective at clearing the virus while maintaining graft function in both kidney alone and simultaneous kidney-pancreas transplant recipients. However, there is a lack of published data on the prevalence and outcomes in simultaneous liver-kidney (SLK) transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* SLK recipients transplanted at MDMC between 2015-2020

Exclusion Criteria:

* Below 18 years of age
* Patients who did not undergo SLK transplant at MDMC

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: SLK transplant recipients who were transplanted at MDMC over a 6-year period (2015 to 2020).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-11-17 (Estimated); Study Completion 2022-11-17 (Estimated)

PRIMARY OUTCOMES:
To characterize the prevalence of BKV in the SLK patient population at MDMC. | over a 6-year period (2015 to 2020).
  number of SLK transplant recipients who were transplanted at MDMC

CONTACTS AND LOCATIONS:
Overall Officials: Lori Kautzman, MD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Kotton CN, Kamar N, Wojciechowski D, Eder M, Hopfer H, Randhawa P, Sester M, Comoli P, Tedesco Silva H, Knoll G, Brennan DC, Trofe-Clark J, Pape L, Axelrod D, Kiberd B, Wong G, Hirsch HH; Transplantation Society International BK Polyomavirus Consensus Group. The Second International Consensus Guidelines on the Management of BK Polyomavirus in Kidney Transplantation. Transplantation. 2024 Sep 1;108(9):1834-1866. doi: 10.1097/TP.0000000000004976. Epub 2024 Apr 12. PMID 38605438